CLINICAL TRIAL: NCT03336619
Title: A Phase III, Randomized, Double-Blind, Placebo Controlled Trial to Evaluate the Efficacy and Safety of Nitazoxanide in the Treatment of Uncomplicated Influenza
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Romark Laboratories L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RM08-3004
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Results first posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-04

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — nitazoxanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nitazoxanide (Active Comparator): Two Nitazoxanide 300 mg tablets orally twice daily (b.i.d.) for 5 days
  Interventions: Drug: Nitazoxanide
- Placebo (Placebo Comparator): Two Placebo tablets orally twice daily (b.i.d.) for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitazoxanide — Nitazoxanide 600 mg administered orally twice daily for five days
  Other Names: NTZ; NT-300
  Arms: Nitazoxanide
Drug: Placebo — Placebo administered orally twice daily for five days
  Arms: Placebo

SUMMARY:
Trial to evaluate efficacy and safety of nitazoxanide (NTZ) in the treatment of uncomplicated influenza.

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, placebo controlled trial to evaluate efficacy and safety of nitazoxanide (NTZ) in the treatment of uncomplicated influenza.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects at least 12 years of age
2. Presence of clinical signs and/or symptoms consistent with an acute illness compatible with influenza infection (each of the following is required):

   1. oral temperature ≥99.4°F or ≥37.4°C (obtained in office or self- measured within 12 hours prior to screening - if self-measured, subjects must also have taken an antipyretic within 4 hours prior to screening), AND
   2. at least one of the following respiratory symptoms (cough, sore throat, nasal obstruction), AND
   3. one of the following constitutional symptoms (fatigue, headache, myalgia, feverishness).
3. Confirmation of influenza A or B infection in the local community by one of the following means:

   1. the institution's local laboratory,
   2. the local public health system,
   3. the national public health system, OR
   4. a laboratory of a recognized national or multinational influenza surveillance scheme.
4. Onset of illness no more than 40 hours before enrollment in the trial.

   Note: Time of onset of illness is defined as either the earlier of:
   1. the time when the temperature was first measured as elevated, OR
   2. the time when the subject experienced the presence of at least one respiratory symptom AND the presence of at least one constitutional symptom.
5. Willing and able to provide written informed consent (including assent by legal guardian if under 18 years of age) and comply with the requirements of the protocol, including completion of the patient diary.

Exclusion Criteria:

1. Severity of illness requiring or anticipated to require in-hospital care.
2. Moderate or severe persistent asthma.
3. Cystic fibrosis in children.
4. Stage III or IV (severe or very severe) chronic obstructive pulmonary disease (COPD).
5. Class III or IV congestive heart failure (at least marked limitation of physical activity in which minimal ordinary activity results in fatigue, palpitation, dyspnea, or angina pain)
6. Arrhythmia
7. Immunosuppressive disorders or who are receiving immunosuppressive therapy (e.g., for organ or bone marrow transplants)
8. Untreated HIV infection or treated HIV infection with a CD4 count below 350 cells/mm3 in the last 6 months
9. Persons with sickle cell anemia or other hemoglobinopathies
10. Poorly controlled insulin-dependent diabetes mellitus (HBA1C > 8%)
11. Residents of any age of nursing homes or other long-term care institutions
12. Concurrent infection at the screening examination that requires systemic antimicrobial therapy.
13. Females of childbearing potential who are either pregnant, breast-feeding or are sexually active without the use of birth control. Female subjects of child-bearing potential that are sexually active must have a negative baseline pregnancy test and must agree to continue an acceptable method of birth control for the duration of the study and for 1 month post- treatment. A double barrier method, oral birth control pills administered for at least 2 monthly cycles prior to study drug administration, an IUD, or medroxyprogesterone acetate administered intramuscularly for a minimum of one month prior to study drug administration are acceptable methods of birth control for inclusion into the study. Female subjects are considered of childbearing potential unless they are postmenopausal (absence of menstrual bleeding for 1 year - or 6 months if laboratory confirmation of hormonal status), or have had a hysterectomy, bilateral tubular ligation or bilateral oophorectomy.
14. Receipt of any dose of NTZ, oseltamivir, zanamivir, peramivir, laninamivir, baloxavir, amantadine or rimantadine within 3 days prior to screening.
15. Prior treatment with any investigational drug therapy within 30 days prior to screening.
16. Subjects with active respiratory allergies or subjects expected to require anti-allergy medications during the study period for respiratory allergies.
17. Known sensitivity to NTZ or any of the excipients comprising the NTZ tablets.
18. Subjects unable to take oral medications.
19. Presence of any pre-existing illness that, in the opinion of the Investigator, would place the subject at an unreasonably increased risk through participation in this study.
20. Subjects who, in the judgment of the Investigator, will be unlikely to comply with the requirements of this protocol.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1030 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Rossignol, M.D., Ph.D., Study Director — Romark Laboratories L.C.
Locations (35):
- United States (31):
  - Vanguard Study Site, Alabaster, Alabama
  - Vanguard Study Site, Birmingham, Alabama
  - Vanguard Study Site, Hoover, Alabama
  - Vanguard Study Site, Pelham, Alabama
  - Vanguard Study Site, Goodyear, Arizona
  - Vanguard Study Site, Tolleson, Arizona
  - Vanguard Study Site, Hot Springs, Arkansas
  - Vanguard Study Site, Anaheim, California
  - Vanguard Study Site, Westminster, California
  - Vanguard Study Site, Lauderdale Lakes, Florida
  - Vanguard Study Site, Orlando, Florida
  - Vanguard Study Site, Valparaiso, Indiana
  - Vanguard Study Site, New Orleans, Louisiana
  - Vanguard Study Site, St Louis, Missouri
  - Vanguard Study Site, Missoula, Montana
  - Vanguard Study Site, Brooklyn, New York
  - Vanguard Study Site, Cincinnati, Ohio
  - Vanguard Study Site, Columbus, Ohio
  - Vanguard Study Site, Dayton, Ohio
  - Vanguard Study Site, Medford, Oregon
  - Vanguard Study Site, Rapid City, South Dakota
  - Vanguard Study Site, Jackson, Tennessee
  - Vanguard Study Site, Smyrna, Tennessee
  - Vanguard Study Site, Austin, Texas
  - Vanguard Study Site, Carrollton, Texas
  - Vanguard Study Site, Dallas, Texas
  - Vanguard Study Site, Fort Worth, Texas
  - Vanguard Study Site, Houston, Texas
  - Vanguard Study Site, Pharr, Texas
  - Vanguard Study Site, Plano, Texas
  - Vanguard Study Site, St. George, Utah
- Australia (3):
  - Vanguard Study Site, Morayfield, Queensland
  - Vanguard Study Site, Sherwood, Queensland
  - Vanguard Study Site, Victoria Point, Queensland
- Vanguard Study Site, Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nitazoxanide | Placebo
Started | 515 | 515
Positive for Influenza by RT-PCR at Baseline (Intent-to-treat Infected [ITTI] Population) | 314 | 306
Completed | 301 | 290
Not Completed | 214 | 225
Not completed — Completed Study, but not positive for influenza by RT-PCR (not included in ITTI population) | 192 | 204
Not completed — Withdrawal by Subject | 17 | 16
Not completed — Adverse Event | 2 | 5
Not completed — Physician Decision | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitazoxanide | Placebo | Total
Number analyzed (Participants) | 515 | 515 | 1030
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.0 (15.11) | 36.3 (16.14) | 35.6 (15.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 292 | 285 | 577
  Male | 223 | 230 | 453
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 47 | 54 | 101
  Hispanic | 194 | 194 | 388
  White | 256 | 260 | 516
  Other | 18 | 7 | 25
Weight [Mean (Standard Deviation); unit: kg] | 83.1 (24.28) | 81.2 (22.58) | 82.1 (23.45)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.6 (7.85) | 29.1 (7.27) | 29.3 (7.57)
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 53 | 49 | 102
  Past Smoker | 64 | 69 | 133
  Never Smoked | 398 | 397 | 795
Time from Onset of Symptoms at First Study Drug Intake (ITTI) [Mean (Standard Deviation); unit: hours] — Population: The Intent-to-Treat-Infected (ITTI, primary efficacy) population consisted of all subjects positive for influenza at Baseline.
  hours
    number analyzed (Participants) | 314 | 306 | 620
    (all) | 26.0 (9.0) | 26.5 (8.2) | 26.2 (8.6)
Presence of Anti-Influenza Antibodies at Baseline [Count of Participants; unit: Participants] — Population: Analysis population consists of subjects positive for influenza infection at Baseline who had Baseline serology samples available for detection of anti-influenza antibodies.
  Participants
    number analyzed (Participants) | 297 | 286 | 583
    Anti-Influenza Antibodies Detected at Baseline | 188 | 181 | 369
    Anti-Influenza Antibodies Not Detected at Baseline | 109 | 105 | 214

OUTCOME MEASURES:

1. Primary Outcome: Time From First Dose to Symptom Response
Description: Subjects used the FLU-PRO questionnaire once daily in the evening to score the severity of 32 FLU-PRO symptoms. Symptom response was deemed achieved when the rating for each of the 32 FLU-PRO symptoms was ≤ its assigned threshold for 2 consecutive daily diary periods without use of symptom relief medication. The symptom response thresholds were developed by applying an algorithm to blinded symptoms data to select the set of 32 symptom thresholds most closely associated with patient-reported usual health.
Time Frame: Up to 21 days
Population: The ITTI (primary efficacy) population consisted of all subjects positive for influenza by RT-PCR at Baseline.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 314 | 306
hours | 155.1 [103.7 to 266.3] | 153.9 [100.2 to 270.7]
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.3765, Gehan-Wilcoxon; Analysis used a Gehan-Wilcoxon test stratified by time from symptom onset at enrollment and influenza vaccination status

2. Secondary Outcome: Time From First Dose to Ability to Perform All Normal Activities
Description: Subjects completed a diary including rating ability to perform normal activities on a scale from 0 (able to perform no normal activities) to 10 (able to perform all normal activities) daily in the evening. The time from first dose to ability to perform all normal activities is the time in hours between the first dose of study medication and that time when the subject first reported a score of "10" (able to perform all normal activities) for two consecutive daily diary periods without use of symptom relief medication.
Time Frame: Up to 21 days
Population: The ITTI (primary efficacy) population consisted of all subjects positive for influenza by RT-PCR at Baseline.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 314 | 306
hours | 201.8 [126.6 to 362.7] | 200.8 [127.5 to 347.2]
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.6331, Gehan-Wilcoxon; Gehan-Wilcoxon test stratified by time from symptom onset at enrollment and influenza vaccination status

3. Secondary Outcome: Number of Subjects Experiencing One or More Complications of Influenza
Description: Complications of influenza infection included pneumonia, otitis media, bronchitis, sinusitis, worsening of pre-existing health conditions, systemic antibiotic use for infections secondary to influenza infection, hospitalization due to influenza or complications of influenza and death.
Time Frame: Up to 21 days
Population: The ITTI (primary efficacy) population consisted of all subjects positive for influenza by RT-PCR at Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 314 | 306
Participants | 50 | 45
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.7382, Fisher Exact

4. Secondary Outcome: Time to Symptom Response Excluding the FLU-PRO Gastrointestinal and Eye Domains
Description: Subjects used the FLU-PRO questionnaire once daily in the evening to score the severity of 32 FLU-PRO symptoms. Symptom response was deemed achieved when the rating for each of the 25 FLU-PRO symptoms (excluding gastrointestinal and eye symptoms) was ≤ its assigned threshold for 2 consecutive daily diary periods without use of symptom relief medication. The symptom response thresholds were developed by applying an algorithm to blinded symptoms data to select the set of 25 symptom thresholds most closely associated with patient-reported usual health.
Time Frame: Up to 21 days
Population: The ITTI (primary efficacy) population consisted of all subjects positive for influenza by RT-PCR at Baseline
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 314 | 306
hours | 152.2 [100.8 to 248.9] | 151.7 [97.8 to 268.7]
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.3236, Gehan-Wilcoxon; Gehan-Wilcoxon test stratified by time from symptom onset to enrollment and influenza vaccination status

5. Other Pre Specified Outcome: Time to Return to Usual Health
Description: Subjects completed the FLU-PRO questionnaire including global assessment questions daily in the evening. The time from first dose to ability to return to usual health is the time in hours from the first dose of study medication to the first time when the subject answered "Have you returned to your usual health?" with "yes" for two consecutive daily diary periods without the use of symptom relief medication.
Time Frame: 21 days
Population: The ITTI (primary efficacy) population consisted of all subjects positive for influenza by RT-PCR at Baseline.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 314 | 306
hours | 176.6 [120.0 to 315.0] | 202.1 [126.6 to 322.1]
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.0483, Gehan-Wilcoxon; Gehan-Wilcoxon test stratified by time from symptom onset at enrollment and influenza vaccination status

6. Other Pre Specified Outcome: Proportion of Diaries Misclassified by Novel Response Definition
Description: The proportion of patient diaries misclassified by the response definition used for the primary efficacy analysis compared to patient reported usual health. A diary was considered "misclassified" if the response definition predicted "responded" and the patient reported not being at usual health or if the response definition predicted "not responded" and the patient reported being at usual health.
Time Frame: 21 days
Population: The ITTI (primary efficacy) population consisted of all subjects positive for influenza by RT-PCR at Baseline. Per the Statistical Analysis Plan, the response definition misclassification rate was to be calculated prior to unblinding including all data for subjects in the ITTI population.
Measure: Number; unit: diaries
Units Other Than Participants: Diaries
Groups:
- ITTI Population: The ITTI (primary efficacy) population consisted of all subjects positive for influenza by RT-PCR at Baseline.
Arm/Group | ITTI Population
Number analyzed (Participants) | 620
Number analyzed (Diaries) | 396128
diaries | 0.20131

7. Post Hoc Outcome: Correlation Coefficient for Sustained Response and Return to Usual Health
Description: The correlation coefficient between sustained response and return to usual health was calculated for the pooled ITTI population (i.e., not by treatment group) as a measure of association between the primary endpoint response definition and its intended anchor, patient-reported return to usual health.
Time Frame: 21 days
Population: The correlation coefficient between sustained response and return to usual health was to be calculated prior to unblinding including all data for subjects in the ITTI population, consistent with the misclassification rate as specified in the statistical analysis plan.
Measure: Number; unit: correlation coefficient
Arm/Group | ITTI Population
Number analyzed (Participants) | 620
correlation coefficient | 0.51

8. Post Hoc Outcome: Time to Return to Usual Health, Placebo-Treated Subjects by Baseline Antibody Status
Description: Survival analysis of Time to Return to Usual Health was repeated for subjects with laboratory-confirmed influenza (ITTI population) who were randomized to the placebo treatment group by whether the subjects had detectable anti-influenza antibodies at Baseline.
Time Frame: 21 days
Population: Subjects with laboratory-confirmed influenza (ITTI population) who were randomized to the placebo treatment group by whether the subjects had detectable anti-influenza antibodies at Baseline.
Measure: Median (Inter-Quartile Range); unit: hours
Groups:
- Placebo-Treated Subjects With Detectable Antibodies at Baseline: Subjects with laboratory-confirmed influenza (ITTI population) randomized to receive placebo who had anti-influenza antibodies detected in a Baseline serum sample.
- Placebo-Treated Subjects Without Detectable Antibodies at Baseline: Subjects with laboratory-confirmed influenza (ITTI population) randomized to receive placebo who had no anti-influenza antibodies detected in a Baseline serum sample.
Arm/Group | Placebo-Treated Subjects With Detectable Antibodies at Baseline | Placebo-Treated Subjects Without Detectable Antibodies at Baseline
Number analyzed (Participants) | 180 | 104
hours | 224.1 [128 to 359] | 261.5 [162 to 504]

9. Post Hoc Outcome: Time to Sustained Clinical Recovery
Description: Alternative means of endpoint construction were pursued to strengthen the relationship between symptoms-based endpoint measures and subject global assessments of health. Time to Sustained Clinical Recovery is an endpoint based on evidence of meaningful within-subject change sustained for the duration of the study. Time to Sustained Clinical Recovery is the time in hours from the first dose of study medication to the first time at which the subject reports a decrease in total FLU-PRO score from the previous diary with assessment that symptoms are at least "somewhat better than yesterday", no oral temperature ≥100.4 F in the prior 24 hours, and no future increase in any of the FLU-PRO domains except within validated background levels.
Time Frame: 21 days
Population: The ITTI (primary efficacy) population consisted of all subjects positive for influenza by RT-PCR at Baseline.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 314 | 306
hours | 172.2 [81 to 346] | 176.4 [82 to 347]

10. Post Hoc Outcome: Time to Sustained Clinical Recovery by Antibody Status, Placebo-Treated Subjects
Description: as for outcome 9
Time Frame: 21 days
Population: Placebo-treated subjects with and without anti-influenza antibodies detected at Baseline who were positive for influenza by RT-PCR.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Placebo-Treated Subjects With Detectable Antibodies at Baseline | Placebo-Treated Subjects Without Detectable Antibodies at Baseline
Number analyzed (Participants) | 181 | 104
hours | 141.0 [80 to 281] | 247.0 [104 to 457]

11. Post Hoc Outcome: Time to Sustained Clinical Recovery, Subjects Without Detectable Antibodies at Baseline
Description: as for outcome 9
Time Frame: 21 days
Population: Subjects positive for influenza by RT-PCR at Baseline with anti-influenza antibodies detected in a Baseline serum sample.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 109 | 104
hours | 175.4 [84 to 321] | 247.0 [104 to 457]

12. Post Hoc Outcome: Time to Sustained Clinical Recovery, mITTI Population Without Detectable Antibodies at Baseline
Description: as for outcome 9
Time Frame: 21 days
Population: Modified ITTI population consists of subjects with laboratory-confirmed influenza infection without detectable anti-influenza antibodies at Baseline and Baseline subject-reported assessment that symptoms are present, the symptoms are not consistent with the subject's usual health, the symptoms interfere with daily activities, and the symptoms have worsened or remained the same relative to the previous day. Assessment was completed via the Baseline FLU-PRO questionnaire.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 94 | 83
hours | 170.3 [80 to 292] | 263.8 [121 to 462]

ADVERSE EVENTS:
Time Frame: 21 dats
Arm/Group | Nitazoxanide | Placebo
All-Cause Mortality (participants affected / at risk) | 1/515 | 0/515
Serious Adverse Events (participants affected / at risk) | 2/515 | 1/515
Other Adverse Events (participants affected / at risk) | 107/515 | 36/515
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitazoxanide (N=515) | Placebo (N=515)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Typhus (Infections and infestations) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitazoxanide (N=515) | Placebo (N=515)
Diarrhoea (Gastrointestinal disorders) | 34 (41) | 25 (26)
Chromaturia (Renal and urinary disorders) | 75 (75) | 5 (5)
Nausea (Gastrointestinal disorders) | 8 (8) | 13 (13)

LIMITATIONS AND CAVEATS:
Limitations of this study include inability to establish meaningfulness of the novel primary endpoint and selection of patients for whom the benefit of antiviral therapy may be marginal (e.g., vaccinated, antibody-positive, and subjects with improving illness at Baseline).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT03336619/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT03336619/SAP_001.pdf